CLINICAL TRIAL: NCT02457702
Title: Mitochondrial Function in Patients With Severe Liver Disease
Acronym: SLDglyc
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit. Only 2 subjects completed.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jeffrey Browning, PROFESSOR & CHAIR, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU 022015-085; R01DK099289 (NIH)
Record Dates: First submitted 2015-04-30; First posted 2015-05-29 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Hepatic Insufficiency; Hypoalbuminemia
MeSH Terms: conditions — Hepatic Insufficiency; Hypoalbuminemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Orally administered Labeled Glycerol (Experimental): Patients will receive an oral mixture of [U-13C3]glycerol (25 mg/kg) plus unlabeled glycerol (25 mg/kg). The total dose of glycerol will be 50 mg/kg in 100 milliliters of water.
  Interventions: Other: Orally administered labeled glycerol

INTERVENTIONS:
Other: Orally administered labeled glycerol — Oral administration of labeled glycerol

SUMMARY:
The researchers will recruit patients with liver disease at Parkland Hospital. Patients will fast overnight, and the next morning will receive an oral mixture of [U-13C3]glycerol (25 mg/kg) plus unlabeled glycerol (25 mg/kg). The total dose of glycerol will be 50 mg/kg in 100 milliliters of water. The taste is slightly sweet. Blood will be drawn at 60 min and 120 min after the ingestion. Blood glucose will be isolated and analyzed by NMR. The presence of [5,6-13C2]- and [4,5-13C2]glucose indicates preserved mitochondrial function. The researchers anticipate that patients with severe liver disease will show a decrease in mitochondrial function and will inform biosynthetic function of liver mitochondria.

After the first 6 successful exams (see power analysis, below), healthy volunteers (age-, gender-, and race-matched) will be studied at the AIRC and subject to the same protocol.

DETAILED DESCRIPTION:
The researchers will recruit patients with severe liver disease at Parkland Hospital where the procedure will be performed. Age-, gender- and race-matched healthy subjects will be recruited from general population, and the procedure will be performed at the procedure room of the AIRC. Patients at Parkland will be screened and selected by Dr. Jeffrey Browning and Dr. Rodney Infante. After ingestion of 25 mg/kg [U-13C3]glycerol plus 25 mg/kg unlabeled glycerol in water (total glycerol dose, 50 mg/kg), blood will be drawn at +60 and +120 min.

Healthy subjects will make two visits to the AIRC for screening and study procedures. The screening visit will take an hour and the study visit will take 3 hours. Volunteers will be made comfortable in the procedure room of the Research Center. All the study procedures at both Parkland and AIRC will be under the direction of the principal investigator, Dr. Jeffrey Browning.

ELIGIBILITY:
Inclusion Criteria:

* Severe liver disease defined as known liver disease plus at least one of the following: serum albumin less than 3.0 g/dL or INR more than 2.0.

Exclusion Criteria:

* Portal systemic encephalopathy
* Pregnancy or breastfeeding.
* Anemia (hematocrit < 32%)
* Significant weight loss or use of diet pills within previous 6 months.
* Cannot give informed consent, understand the protocol, or tolerate any aspect of the protocol.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-10; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Detection of 13C in plasma glucose by NMR of a blood sample | At 60 minutes and 120 minutes post ingestion
  Once at 60 minutes post ingestion and once at 120 minutes ingestion for a total ot 2 times

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center - Advanced Imaging Research Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No